CLINICAL TRIAL: NCT06190405
Title: Universal Hemoglobin A1c Versus Risk-based Screening for Early Gestational Diabetes Mellitus (EARLY GDM): A Randomized Controlled Trial
Acronym: EARLYGDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Rodney McLaren, Jr., Assistant Professor, Obstetrics and Gynecology, Director of MFM Outpatient Care, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: iRISID-2023-1750
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes; Large for Gestational Age
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal hemoglobin A1c (Experimental): Patients at <16 weeks will have a hemoglobin A1c obtained
  Interventions: Diagnostic Test: Hemoglobin A1c
- Risk-based screening by ACOG with two-step GTT (Active Comparator): Patients at <16 weeks will be assessed for risk factors for diabetes as described by ACOG. If patients meet criteria, they will be screened with two-step screening for gestational diabetes. If patients do not meet criteria, they will not be screened until the routine timing of screening for gestational diabetes.
  Interventions: Diagnostic Test: Risk-based screening by ACOG with two-step GTT

INTERVENTIONS:
Diagnostic Test: Hemoglobin A1c — Patients with a HbA1c <5.7% will be considered a normal test, and they will continue their routine prenatal care, including GDM screening at 24-28 weeks. Patients with a HbA1c ≥5.7% and ≤6.4% will be diagnosed with early GDM. Patients with a HbA1c ≥6.5% will be diagnosed with pregestational diabetes. Patient diagnosed with early GDM or pregestational diabetes will be treated as per usual clinical protocol for gestational/pregestational diabetes.
  Arms: Universal hemoglobin A1c
Diagnostic Test: Risk-based screening by ACOG with two-step GTT — Patients will be assessed for risk factors for GDM as per ACOG. Patients with a negative screen will continue routine care, including GDM screening at 24-28 weeks. Patients with a positive screen will undergo a two-step GTT screening. Patients with a 1-h GTT <135 mg/dL will continue with routine care, including GDM screening at 24-28 weeks. Patients with a 1-h GTT ≥185 mg/dL and <200 mg/dL will be diagnosed with early GDM. Patients with a 1-h GTT ≥200 mg/dL will be diagnosed with pregestational DM. Patients with a 1-h GTT ≥135 mg/dL and <185 mg/dL will undergo a fasting 3-h GTT. Patient will be diagnosed with early GDM by Carpenter and Coustan criteria. Patients will be diagnosed with pregestational DM if their fasting glucose value is ≥126 mg/dL. If patients pass the 3-h GTT, they will continue routine care, including GDM screen at 24-28 weeks with a 3-h GTT. Patient diagnosed with early GDM/pregestational DM will be treated as per usual clinical protocol for GDM/pregestational DM.
  Arms: Risk-based screening by ACOG with two-step GTT

SUMMARY:
The goal of this randomized controlled trial is to compare the rate of large-for-gestational-age neonates between universal screening with glycated hemoglobin (A1C) and early risk-based screening with a glucose tolerance test (GTT) among pregnancies that present to prenatal care at <16 weeks 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to prenatal care ≤16 6/7 weeks of gestation
* Intend to deliver at TJUH

Exclusion Criteria:

* Multifetal gestation
* Pre-pregnancy diagnosis of diabetes mellitus
* History of malabsorptive gastric bypass surgery
* Hemoglobinopathy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 770 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Large-for-gestational age | At time of delivery
  Birthweight ≥90th percentile

SECONDARY OUTCOMES:
Preterm birth | At time of delivery
Stillbirth | At time of delivery
  Fetal death prior to delivery
Shoulder dystocia | At time of delivery
Birth injury | At time of delivery
Neonatal hypoglycemia | From 0 to 24 hours after birth
Neonatal death | 28 days after birth
  Neonatal death within 28 days of birth
Rate of early GDM diagnosis | At time of delivery
Rate of GDM diagnosis after 24 weeks | At time of delivery
Rate of pregestational diabetes | At time of delivery
Rate of patients requiring medication | At time of delivery
  Patients requiring oral hypoglycemic medication and/or insulin treatment
Rate of hypertensive disorders of pregnancy | At time of delivery
  Gestational hypertension and/or preeclampsia